CLINICAL TRIAL: NCT00834496
Title: Sirolimus Switching From Calcinurin Inhibitors (CNI) 90 - 180 Days After Liver Transplantation
Brief Title: Switching From One Type of Anti-rejection Drug (Tacrolimus or Cyclosporine) to Another (Sirolimus) Approximately 90-180 Days After Liver Transplantation
Status: Withdrawn | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 08D.12
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Side Effects of Calcineurin Inhibitors; Renal Toxicity; Hepatic Fibrosis on Biopsy; Neurotoxicity; Post Transplant Diabetes
MeSH Terms: conditions — Neurotoxicity Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Our experience with the use of Sirolimus is delineated below. About 15% to 20% of our patients are currently switched to Sirolimus.Indications for conversion from calcinurin inhibitors (CNIs) to Sirolimus more than 90 days post liver transplantation include:
  * CNI renal toxicity.
  * Hepatic fibrosis on biopsy.
  * CNI neurologic toxicity.
  * Post transplant diabetes. Any of the above 4 indications makes a patient a candidate for conversion from CNIs to Sirolimus at or > 90 days after liver transplantation.
  Interventions: Procedure: Liver biopsy

INTERVENTIONS:
Procedure: Liver biopsy — percutaneous liver biopsy

SUMMARY:
Sirolimus can be safely switched as early as 90 days after liver transplantation with excellent tolerability and amelioration of the calcineurin inhibitor toxicity that initiated the switch.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (18 years or older) patients undergoing liver transplantation at Thomas Jefferson University Hospital.
2. Diagnosed with at least one of the following CNI side effects 90-180 days post transplantation:

   1. CNI renal toxicity. Any liver transplant recipient who has elevated creatinine level (greater than 1.4 mg/dl) and impaired creatinine clearance (MDRD) of 40-60 ml/minute or decreased by 15% compared to baseline in the setting of having a therapeutic CNI level, without suspicion of acute or chronic allograft rejection.
   2. Hepatic fibrosis on biopsy. Any patient who has fibrosis seen on liver biopsy with LFT's 2 times the upper normal limit.
   3. CNI neurologic toxicity. Any patient who has significant neurological side effects from CNIs. This will include the following: seizures not secondary to an epileptogenic focus or any metabolic derangement; alteration of speech ranging from aphasia to slurred speech; inability to be awake and alert.
   4. Post transplant diabetes. Any patient who has developed diabetes after transplant and in whom CNIs are thought to be contributing to poor glycemic control.
3. Signed informed consent at approximately 90 -180 days post transplantation.

Exclusion Criteria:

1. Invasive/surgical therapy within 2 weeks of the 90-180 day post transplantation conversion. (e.g. patients with T-tubes would not be eligible for the study because the T-tube removal will coincide with the conversion date).
2. Open surgical wound at 90-180 days post transplantation.
3. Acute cellular rejection during the first 90-180 days post transplantation.
4. Re-transplants or multiple-organ transplants.
5. Active infection.
6. Pregnancy.
7. Malignancy within 3 years prior to liver transplantation (except adequately treated basal cell carcinoma). Patients with HCC prior to transplant will not be excluded.
8. Total cholesterol >300 mg/dl on medical treatment or triglycerides >150 mg/dl at 90-180 days post transplantation.
9. White blood cell count <3,000/mm3 or platelet count <100,000/mm3 at 90-180 days post transplantation.
10. Ascites.
11. Patients on chemotherapy.
12. Urine protein/creatinine ration > 0.5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: post liver transplant patients taking calcineurin inhibitors (tacrolimus or cyclosporine) as anti-reject medication
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
The primary objective is that acute cellular rejection following a switch to sirolimus will be comparable to the historical rate at our center under calcineurin inhibitors of around 5% for post liver transplant recipients. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Cataldo Doria, MD, PhD, Principal Investigator — Thomas Jefferson University and Hospital
Locations (1):
- THomas Jefferson University and Hospital, Philadelphia, Pennsylvania, United States